CLINICAL TRIAL: NCT06032754
Title: PortoSinusoidal Vascular Diseases and Systemic Sclerosis
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: MVPScS
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-03

CONDITIONS: PSVD With or Without SSc
Keywords: Porto-Sinusoidal Vascular Disease; Nodular regenerative hyperplasia; Systemic sclerosis
MeSH Terms: conditions — Idiopathic Noncirrhotic Portal Hypertension; Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- First group : SSC with PSVD: medical file analysis of patients affected by SSC and PSVD
- Second group : PSVD without SSC: medical file analysis of patients affected by PSVD only
- Third group : SSC without PSVD: medical file analysis of patients affected by SSC only

SUMMARY:
Porto-Sinusoidal Vascular Disorders (PSVD) is a heterogeneous clinico-pathological entity characterized by alterations in small liver vessels. "Nodular regenerative hyperplasia (NRH)" is the most common PSVD. The most frequent liver disease associated with Systemic sclerosis (SSc) is primary biliary cholangitis reported in 2 to 22% of cases. NRH prevalence estimated to 1.4%, may be underestimated as NRH diagnosis is histologic and usually suspected in case of complications due to portal hypertension. Few data are available about NRH associated with SSc resulting in a lack of knowledge of the characteristics and outcome of these patients.

DETAILED DESCRIPTION:
The study aims to compare the outcome of patients with MVPS associated with SSc to patients with MVPS without SSc. This work is a multicenter retrospective study comparing two groups of adult patients, one with MVPS associated with SSc and the other with MVPS without SSc. Patients with MVPS associated with SSc will be recruited from French university hospital departments of Hepatogastroenterology and Internal Medecine. Patients with MVPS without SSc will be recruited from the Beaujon Hospital database dedicated to liver vascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* PSVD (Valdig criteria)
* SSC (ACR/EULAR 2013 criteria)

Exclusion Criteria:

* Liver cirrhosis
* Limited scleroderma
* Autoimmune hepatitis
* Primary biliary cholangitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 3 types of patients : PSVD with SSC, PSVD without SSC, SSC without PSVD will be compared.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Prognosis | 2 years
  To compare prognosis of PSVD patients with or without SSc (less or more gastrointestinal bleeding/portal vein thrombosis)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Caen, Caen, Calvados, France